CLINICAL TRIAL: NCT05198570
Title: Pharmacokinetics of Intravenous Acyclovir in Children Undergoing Hematopoietic Stem Cell Transplantation or High-intensity Antineoplastic Chemotherapy
Brief Title: Pharmacokinetics of Intravenous Acyclovir in Oncologic Paediatric Patients
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Associate Professor of Pharmacology, University of Pisa
Other Study IDs: RC_10/20
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Herpesviridae Infections; Herpes Simplex 1; Varicella Zoster Virus Infection; Transplantation Infection; Oncology
Keywords: Hematopoietic stem cell transplantation; Herpes virus infections; Aciclovir; Children; Pharmacokinetics
MeSH Terms: conditions — Herpesviridae Infections; Varicella Zoster Virus Infection; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravenous Aciclovir: Patients receiving intravenous aciclovir for prophylaxis or treatment of herpes virus infections
  Interventions: Other: Pharmacokinetic analysis
- Oral Aciclovir: Patients receiving oral aciclovir/valaciclovir for prophylaxis or treatment of herpes virus infections
  Interventions: Other: Pharmacokinetic analysis

INTERVENTIONS:
Other: Pharmacokinetic analysis — Population pharmacokinetic analysis of plasma concentrations of aciclovir obtained during routine therapeutic drug monitoring

SUMMARY:
* Herpesvirus infections may be severe in immunocompromised patients, with a high risk of complications and mortality.
* Recipients of hematopoietic stem cell transplant (HSCT) or patients receiving high-intensity chemotherapy for hematological malignancies are the most vulnerable individuals.
* Although the worldwide prevalence of herpes simplex virus 1 (HSV-1) and varicella-zoster virus (VZV), antiviral prophylaxis in seropositive HSCT recipients has significantly reduced the rate of infection.
* Acyclovir (ACV) is the first-choice drug for the prophylaxis or the therapy of that kind of infection.
* Since the beginning, ACV has demonstrated to be characterized by a large interpatient variability, especially in children.
* Therefore, therapeutic drug monitoring and pharmacokinetic studies may help in optimizing drug in children with malignancies.

DETAILED DESCRIPTION:
Herpesvirus infections may lead to severe disease with a high risk of complications and mortality in hematopoietic stem cell transplant (HSCT) recipients, or in patients receiving high-intensity chemotherapy for hematological malignancies. That risk is mainly associated with the worldwide prevalence of herpes simplex virus 1 (HSV-1) that increases consistently with age. In particular, the majority of adult leukemia patients are HSV seropositive, while allogeneic HSCT recipients had post-transplant HSV reactivation. It is worth noting that in the first post-transplant year, symptomatic varicella-zoster virus (VZV) reactivation has a rate of 13% - 55% in adult recipients. Similar percentages of children receiving HSCT had VZV reactivation, being also possible a disseminated infection in 10% of children. However, thanks to antiviral prophylaxis in seropositive HSCT recipients, the rate of infection has significantly dropped.

Among the drugs most used for treatment and prophylaxis of HSV/VZV infections among children who are HSCT recipients or undergo a high-intensity chemotherapy, acyclovir represents the drug of choice. Although its role in preventing and treating herpes virus infections, the pharmacokinetics of acyclovir is highly variable, especially in patients in intensive care units, in those who have organ dysfunction, or in children. In particular, information about the optimal use of acyclovir in children with malignancies is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hematological malignancies
* HSCT recipients who require ACV prophylaxis or treatment for HSV-VZV infection or
* Children undergoing high-intensity antineoplastic chemotherapy who need ACV treatment.
* Intravenous or oral ACV dosing
* Active/available a therapeutic drug monitoring (TDM) protocol for ACV
* Informed consent signed by patient's parents

Exclusion Criteria:

* lack of signed informed consent
* lack of TDM for ACV
* unavailable patient's demographic characteristics

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0-18 years, affected by hematological malignancies, undergoing ACV prophylaxis or treatment for HSV-VZV infection routinely during allogeneic HSCT or ACV treatment during high-intensity chemotherapy, for who a therapeutic drug monitoring (TDM) protocol is available. Patients receive ACV as a standard 1-h intravenous infusion or through the oral administration of valaciclovir
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieve an acyclovir minimum plasma concentration of 0.5 mg/L at steady state | Six months since the beginning of acyclovir administration
  Percentage of patients who achieve an acyclovir minimum plasma concentration at steady state ≥0.5 mg/L, considered as an effective plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Bone Marrow Transplant Unit, Institute for Maternal and Child Health, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No
Individual partecipant data will not be disclosed as per protocol and Ethics Committee requests. Protocol will be shared upon request, as well as the overall findings of the study

REFERENCES:
- [Result] Maximova N, Nistico D, Luci G, Simeone R, Piscianz E, Segat L, Barbi E, Di Paolo A. Population Pharmacokinetics of Intravenous Acyclovir in Oncologic Pediatric Patients. Front Pharmacol. 2022 Apr 14;13:865871. doi: 10.3389/fphar.2022.865871. eCollection 2022. PMID 35496277